CLINICAL TRIAL: NCT05082961
Title: Circulating Immunes Cells, Cytokines and Brain Radiotherapy
Acronym: CYRAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Ligue contre le cancer, France (Other); Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-A01862-39
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- X-ray photon therapy + biological samples (Other)
  Interventions: Other: Collection of blood samples
- Protontherapy + biological samples (Other)
  Interventions: Other: Collection of blood samples

INTERVENTIONS:
Other: Collection of blood samples — Samples to evaluate the circulating CD8+ T cell count.

SUMMARY:
Patients with malignant tumours of the cephalic pole have a poor prognosis, despite a wide range of treatments. prognosis despite a large therapeutic arsenal. Among this arsenal, radiotherapy (RT) is one of the standard treatments for these tumours. However, this treatment can cause damage to the surrounding healthy tissue, has limited efficacy in hypoxic However, this treatment can cause damage to the surrounding healthy tissue, has limited efficacy in hypoxic tissue and can promote pro-tumour inflammation.

In these circumstances, hadrontherapy, which uses charged heavy particles, such as protons or carbon ions, is the preferred treatment. protons or carbon ions, seems more appropriate for the treatment of these tumours. However, although inflammation plays a major role in tumour development and tumour development and therapeutic response, few studies have evaluated the immune response response after proton therapy (PT) and carbon therapy (CT). The objective of this project is to study the effect of hadrontherapy on resident/circulating inflammation after brain irradiation. brain irradiation. In a first step, the impact of different PT and CT TEL on macrophages (MФ), the most abundant immune cells in malignant solid tumours, will be evaluated in vitro. malignant solid tumours, will be evaluated in vitro. In a second step, the evolution of circulating leukocytes after brain irradiation with X-rays or protons will be studied in vivo in rodents and patients. rodent and patient. In this project, we propose to study for the first time the inflammatory response after hadrontherapy in the context of a cephalic tumour. cephalic tumour. These results will allow a better understanding of the biological response response following PT and CT with the aim of optimising RT and potentially and potentially translate these data to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Head and neck cancer: (upper aerodigestive tract, cavum, facial sinus, skull base, brain) operated
* Surgery for complete tumour resection or with microscopic residue R1
* All possible histologies: squamous cell carcinoma, undifferentiated carcinoma of the nasopharyngeal type (UCNT), adenocarcinoma, adenoid cystic carcinoma, chordoma, chondrosarcoma,meningioma other tumours
* Patients undergoing exclusive postoperative radiotherapy with a minimum total dose of 54 Gy of X-ray photon radiation or equivalent proton radiation.
* Patient affiliated to a social security scheme
* Signature of the informed consent before any specific procedure related to the study

Exclusion Criteria:

* Macroscopic postoperative tumour residue R2
* Previous cancer within 5 years (except treated basal cell skin carcinoma and treated cervical cancer).
* Previous radiotherapy (except brachytherapy of the cervix or prostate)
* Chemotherapy or other systemic oncological treatment (cetuximab) concomitant with radiotherapy
* Long-term immunosuppressive or corticosteroid therapy
* Patient deprived of liberty or under guardianship, protected adult
* Patient unable to undergo trial monitoring for geographical, social or psychopathological reasons
* Pregnant or breastfeeding woman
* Emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
CD8+ T-cell count. | up to 3 months

SECONDARY OUTCOMES:
CD4+ Lymphocytes T count | up to 3 months
Regulatory T cells | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thariat J, Pham TN, Coupey J, Clarisse B, Grellard JM, Rousseau N, Cesaire M, Valable S. CYRAD: a translational study assessing immune response to radiotherapy by photons or protons in postoperative head and neck cancer patients through circulating leukocyte subpopulations and cytokine levels. BMC Cancer. 2024 Oct 5;24(1):1230. doi: 10.1186/s12885-024-13002-1. PMID 39369231